CLINICAL TRIAL: NCT01284387
Title: A Phase 2, 24-Month, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Amyloid-Imaging Positron Emission Tomography (PET) and Safety Study of ACC-001 and QS-21 Adjuvant in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Amyloid Imaging And Safety Study Of ACC-001 In Subjects With Mild to Moderate Alzheimer's Disease
Acronym: ACCTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACC-001-ALZ-2001
Record Dates: First submitted 2011-01-20; First posted 2011-01-27 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Alzheimer's Disease
Keywords: Mild to moderate Alzheimer's disease; immunization; amyloid imaging; injection; vaccine
MeSH Terms: conditions — Alzheimer Disease | interventions — vanutide cridificar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3 μg ACC-001 / QS-21 50 μg IM dose 1 (Experimental): 3 μg ACC-001 / QS-21 50 μg IM
  Interventions: Biological: ACC-001 (vanutide cridificar)
- 10 μg ACC-001 / QS-21 50 μg IM dose 2 (Experimental): 10 μg ACC-001 / QS-21 50 μg IM
  Interventions: Biological: ACC-001 (vanutide cridificar)
- Placebo - Phosphate buffered saline (PBS) IM dose (No Intervention): Placebo - Phosphate buffered saline (PBS) IM

INTERVENTIONS:
Biological: ACC-001 (vanutide cridificar) — Comparisons of 2 different doses of ACC-001 or placebo for 24 months
  Other Names: vanutide cridificar
  Arms: 10 μg ACC-001 / QS-21 50 μg IM dose 2; 3 μg ACC-001 / QS-21 50 μg IM dose 1

SUMMARY:
A Phase II clinical research study to evaluate the efficacy and safety of two different dose levels of an injectable investigational treatment (ACC-001) in subjects with Mild-to-Moderate Alzheimer's disease. ACC-001 (vanutide cridificar) is a beta amyloid fragment attached to a carrier protein. It is intended to help induce an antibody response against beta amyloid and is administered as an intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD
* Age from 50 to 89
* Mini-Mental Status Exam score of 18-26 inclusive
* Brain magnetic resonance imaging (MRI) scan consistent with the diagnosis of AD
* Stable doses of medications (cholinesterase inhibitors and memantine allowed)
* Caregiver able to attend all clinic visits with patient
* Amyloid burden on screening PET scan consistent with diagnosis of AD

Exclusion Criteria:

* Significant neurological disease other than AD
* Major psychiatric disorder
* Significant systemic illness
* History of stroke, seizure or autoimmune disease
* History of myocardial infarction within the last 2 years
* Smoking greater than 20 cigarettes per day
* Anticonvulsants, anti-Parkinson's, anticoagulant, or narcotic medications (anticonvulsants used for non-seizure reasons are allowed)
* Prior treatment experimental immunotherapeutics or vaccines for AD
* Women of childbearing potential
* Presence of pacemakers, CSF shunts, or foreign metal objects in the eyes, skin or body

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of ACC-001 in combination with an adjuvant immunostimulatory agent (QS-21), administered intramuscularly compared to placebo on cerebral amyloid burden in subjects with mild to moderate Alzheimer's disease. | 24 Months

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of 2 dosage levels of ACC-001 plus QS-21 vs. placebo in subjects with mild to moderate AD. | 24 Months
  As assessed by:
  * The incidence and severity of treatment-emergent adverse events (TEAEs); and
  * Clinically important changes in safety assessment results (vital signs, weight, clinical laboratory tests, electrocardiograms [ECGs], brain magnetic resonance imaging [MRIs], and physical and neurological examinations).
Exploratory Outcome Measure: To assess the effects of ACC-001 compared to placebo as measured by change from baseline in disease biomarkers. | 24 Months
Exploratory Outcome Measure: To assess the effects of ACC-001 compared to placebo as measured by change from baseline in measurements of immunogenicity. | 24 Months
Exploratory Outcome Measure: To assess the effects of ACC-001 compared to placebo as measured by change from baseline in cognitive and functional scales. | 24 Months
Exploratory Outcome Measure: To assess the effects of ACC-001 compared to placebo as measured by change from baseline in health outcome measures. | 24 Months

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Janssen AI Investigational Site, Sun City, Arizona
  - Janssen AI Investigational Site, La Jolla, California
  - Janssen AI Investigational Site, Long Beach, California
  - Janssen AI Investigational Site, Los Angeles, California
  - Janssen AI Investigational Site, Oxnard, California
  - Janssen AI Investigational Site, San Diego, California
  - Janssen AI Investigational Site, San Francisco, California
  - Janssen AI Investigational Site, Washington D.C., District of Columbia
  - Janssen AI Investigational Site, Miami, Florida
  - Janssen AI Investigational Site, Ocala, Florida
  - Janssen AI Investigational Site, Orlando, Florida
  - Janssen AI Investigational Site, Sunrise, Florida
  - Janssen AI Investigational Site, Tampa, Florida
  - Janssen AI Investigational Site, West Palm Beach, Florida
  - Janssen AI Investigational Site, Scarborough, Maine
  - Janssen AI Investigational Site, Boston, Massachusetts
  - Janssen AI Investigational Site, Kansas City, Missouri
  - Janssen AI Investigational Site, Las Vegas, Nevada
  - Janssen AI Investigational Site, Princeton, New Jersey
  - Janssen AI Investigational Site, Albany, New York
  - Janssen AI Investigational Site, New York, New York
  - Janssen AI Investigational Site, Centerville, Ohio
  - Janssen AI Investigational Site, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Ketter N, Liu E, Di J, Honig LS, Lu M, Novak G, Werth J, LePrince Leterme G, Shadman A, Brashear HR. A Randomized, Double-Blind, Phase 2 Study of the Effects of the Vaccine Vanutide Cridificar with QS-21 Adjuvant on Immunogenicity, Safety and Amyloid Imaging in Patients with Mild to Moderate Alzheimer's Disease. J Prev Alzheimers Dis. 2016;3(4):192-201. doi: 10.14283/jpad.2016.118. PMID 29199321